CLINICAL TRIAL: NCT01401829
Title: Psychosocial Benefits of Exercise in Endometrial Cancer Survivors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to lack of funding required to continue the study.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ROG-SIU-11-004
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; aerobic walking; stretching/flexibility exercises; quality of life
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 75 weekly minutes walking (Experimental): 12-week physical activity intervention group with a goal of 75 minutes of moderate intensity exercise (walking) per week
  Interventions: Behavioral: 75 weekly minutes walking
- 150 weekly minutes walking (Experimental): 12 week physical activity intervention group with a goal of 150 minutes of moderate intensity exercise (walking) per week
  Interventions: Behavioral: 150 weekly minutes walking
- Stretching and Flexibility exercise (Active Comparator): Stretching/Flexibility exercise
  Interventions: Behavioral: Stretching/Flexibility exercise

INTERVENTIONS:
Behavioral: 150 weekly minutes walking — 12 week physical activity intervention group with a goal of 150 minutes of moderate intensity exercise (walking) per week on a treadmill while supervised by exercise specialists who are certified by ACSM and trained and monitored for quality control and safety
  Other Names: moderate intensity aerobic walking
  Arms: 150 weekly minutes walking
Behavioral: 75 weekly minutes walking — 12 week physical activity intervention group with a goal of 75 minutes of moderate intensity exercise (walking) per week on a treadmill while supervised by exercise specialists who are certified by ACSM and trained and monitored for quality control and safety
  Other Names: moderate intensity aerobic walking
  Arms: 75 weekly minutes walking
Behavioral: Stretching/Flexibility exercise — 12 week stretching intervention group with a goal of 3 sessions per week while supervised by exercise specialists who are certified by ACSM and trained and monitored for quality control and safety
  Other Names: stretching exercise
  Arms: Stretching and Flexibility exercise

SUMMARY:
To determine if weekly exercise compared to stretching has an effect on fatigue, depression, and anxiety in endometrial cancer survivors.

DETAILED DESCRIPTION:
Endometrial cancer is the most prevalent gynecologic cancer in women. Because of its excellent 5 year survival rate of 83%, addressing longer term cancer effects in this group is an important aspect of cancer survivor care. Unfortunately, women with a history of endometrial cancer may report persistent levels of fatigue, depression, and anxiety that are, on average, higher than those of healthy, gynecologic out-patients. Physical activity is one potential approach to reducing these symptoms, but little is known about the effects of physical activity in endometrial cancer survivors specifically. Furthermore, current evidence is insufficient to make recommendations regarding the optimal exercise amount, type, and duration for improving fatigue, depression, or anxiety after a cancer diagnosis (any cancer type).

This pilot, randomized trial is unique in its focus on endometrial cancer survivors, a previously understudied population with a large potential for benefiting from regular physical activity. Two separate walking intervention groups will work with an exercise specialist three times a week to walk for either 75 minutes (group 1) or 150 minutes (group 2) weekly. The participants will start out slowly and then gradually increase to the particular group goal of 75 or 150 minutes. The stretching exercise group will work with an exercise specialist doing stretching/flexibility exercises three times a week starting with 15 seconds and then gradually increasing to 30 seconds of holding the stretch.

ELIGIBILITY:
Inclusion Criteria:

* 1) Female, 18 to 70 years of age with history of Stage I, II, or III endometrial cancer diagnosis occurring at least 6 months prior to study enrollment,
* 2) if chemotherapy or radiation therapy was received, patient must be ≥ 4 weeks post final primary treatment administration,
* 3) if patient has undergone surgical procedure, must be ≥ 8 weeks post-procedure or cleared by surgeon for moderate intensity walking,
* 4) English speaking,
* 5) medical clearance for participation provided by primary care physician or oncologist,
* 6) average fatigue over the past week of ≥3 on a 1 to 10 Likert scale or worrying thoughts ≥ a lot of the time or enjoy the things they used to a little/ not at all.

Exclusion Criteria:

* 1) metastatic or recurrent endometrial cancer,
* 2) inability to ambulate without assistance,
* 3) unstable angina,
* 4) New York Heart Association class II, III, or IV congestive heart failure,
* 5) uncontrolled asthma,
* 6) having been told by a physician to only do exercise prescribed by a physician,
* 7) dementia or organic brain syndrome,
* 8) schizophrenia or active psychosis,
* 9) participating, on average, in more than 20 minutes of physical activity on two or more days per week during the past six months,
* 10) anticipates undergoing elective surgery during the duration of the intervention which would interfere with the intervention participation,
* 11) does not live or work less than 50 miles from the study site,
* 12) lack of transportation to the study site,
* 13) plans to move residence out of the local area during the study duration,
* 14) plans to travel out of the local area for more than a week during the intervention,
* 15) contraindication to participation in physical activity,
* 16) non-compliant with sleep apnea treatments.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
fatigue | Change from baseline at 12 weeks
  13-item multi-dimensional fatigue scale [i.e. Fatigue Symptom Inventory (FACT-F)]

SECONDARY OUTCOMES:
Depression and Anxiety | Change from baseline at 8 weeks
  14 item Hospital Anxiety and Depression Scale (PROMIS)
Depression and Anxiety | Change in baseline at 12 weeks
  14 item Hospital Anxiety and Depression Scale (PROMIS)
Task self-efficacy | Change in baseline at 8 weeks
  4 item scale for chronic disease patients
Task self-efficacy | Change in baseline at 12 weeks
  4 item scale for chronic disease patients
Quality of Life | Change in baseline at 8 weeks
  Functional Assessment of Cancer Therapy-Endometrial and the Satisfaction With Life Scale
Quality of Life | Change in baseline at 12 weeks
  Functional Assessment of Cancer Therapy-Endometrial and the Satisfaction With Life Scale
Body Mass Index (BMI) | Change in baseline at 8 weeks
  BMI calculated with weight and height
Body Mass Index (BMI) | Change in baseline at 12 weeks
  BMI calculated with weight and height
Body Composition | Change in baseline at 8 weeks
  Bioelectrical Impedance
Body Composition | Change in baseline at 12 weeks
  Bioelectrical Impedance
Waist and Hip circumferences | Change in baseline at 8 weeks
  the average of three measures of waist and hip (each) using a tape measure
Waist and Hip circumferences | Change in baseline at 12 weeks
  the average of three measures of waist and hip (each) using a tape measure
fitness | Change in baseline at 8 weeks
  submaximal fitness test
fitness | Change in baseline at 12 weeks
  submaximal fitness test
muscle strength | Change in baseline at 8 weeks
  back/leg dynamometer and hand grip dynamometer
muscle strength | Change in baseline at 12 weeks
  back/leg dynamometer and hand grip dynamometer
feasibility | one year
  Number of patients recruited, Number of patients who complete the walking intervention, Number of adverse events reported, and Number of patients who complete the study
demographic, lifestyle, and medical covariates | one year
  self-administered survey

CONTACTS AND LOCATIONS:
Overall Officials: Laura Q. Rogers, MD, MPH, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Background] Rogers LQ. Objective monitoring of physical activity after a cancer diagnosis: challenges and opportunities for enhancing cancer control. Phys Ther Rev. 2010 Jun 1;15(3):224-237. doi: 10.1179/174328810X12814016178872. PMID 21603254
- [Background] Rogers LQ, Markwell S, Hopkins-Price P, Vicari S, Courneya KS, Hoelzer K, Verhulst S. Reduced barriers mediated physical activity maintenance among breast cancer survivors. J Sport Exerc Psychol. 2011 Apr;33(2):235-54. doi: 10.1123/jsep.33.2.235. PMID 21558582
- [Background] Rogers LQ, Hopkins-Price P, Vicari S, Markwell S, Pamenter R, Courneya KS, Hoelzer K, Naritoku C, Edson B, Jones L, Dunnington G, Verhulst S. Physical activity and health outcomes three months after completing a physical activity behavior change intervention: persistent and delayed effects. Cancer Epidemiol Biomarkers Prev. 2009 May;18(5):1410-8. doi: 10.1158/1055-9965.EPI-08-1045. Epub 2009 Apr 21. PMID 19383889
- [Background] Rogers LQ, Malone J, Rao K, Courneya KS, Fogleman A, Tippey A, Markwell SJ, Robbins KT. Exercise preferences among patients with head and neck cancer: prevalence and associations with quality of life, symptom severity, depression, and rural residence. Head Neck. 2009 Aug;31(8):994-1005. doi: 10.1002/hed.21053. PMID 19340875
- [Background] Rogers LQ, Courneya KS, Robbins KT, Rao K, Malone J, Seiz A, Reminger S, Markwell SJ, Burra V. Factors associated with fatigue, sleep, and cognitive function among patients with head and neck cancer. Head Neck. 2008 Oct;30(10):1310-7. doi: 10.1002/hed.20873. PMID 18642320
- [Background] Rogers LQ, Markwell SJ, Courneya KS, McAuley E, Verhulst S. Exercise preference patterns, resources, and environment among rural breast cancer survivors. J Rural Health. 2009 Fall;25(4):388-91. doi: 10.1111/j.1748-0361.2009.00249.x. PMID 19780920
- See also: American Cancer Society — http://www.cancer.org/index
- See also: American College of Sports Medicine — http://www.acsm.org/
- See also: National Cancer Institute of the National Institutes of Health — http://www.cancer.gov/